CLINICAL TRIAL: NCT06516107
Title: Understanding Parental Stress and Quality of Life in Families of Children With Diplegic Cerebral Palsy: Key Influencing Factors
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Alaa Noureldeen Kora, Lecturer at the Department of Physical Therapy for Pediatrics and Pediatric Surgery, Sinai University
Other Study IDs: SU.REC.2024(30H)
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Stress; Diaplegia; Cerebral Palsy
Keywords: Cerebral palsy; Quality of life; Parental stress
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 Group of parents of children with diplegic cerebral palsy: Parents of children between the ages of 2 and 4.8 who had been diagnosed with diplegic CP and were in a stable clinical and medical state will be included in this study. However, parents of children with behavioral problems, a history of ongoing heart disease, a botulinum toxin injection within the six months previous to the study, chronic chest disease, significant visual or auditory impairment, or parents with limited literacy will not allowed to participate in the study

SUMMARY:
PURPOSE:

To estimate the relationships between the child, parents, and family factors and parent stress and QoL among parents of children with diplegic CP.

BACKGROUND:

Cerebral palsy (CP) is considered the primary reason of motor impairment among children worldwide. Compared to parents of typically developing children, parents of children with cerebral palsy (CP) experience higher levels of stress and reduced quality of life (QoL).

HYPOTHESES:

There is no relation between the level of functional impairment among children with diplegic CP and their parental stress and QOL.

RESEARCH QUESTION:

Is there a relationship between the level of functional impairment among children with diplegic CP and the degree of their parental stress and quality of life?

ELIGIBILITY:
Inclusion Criteria:

* Parents of children between the ages of 2 and 4.8 who had been diagnosed with diplegic CP.

  * Parents of children with diplegic CP who were in a stable clinical and medical state.

Exclusion Criteria:

* parents of children with behavioral problem.
* a history of ongoing heart disease
* a botulinum toxin injection within the six months previous to the study
* chronic chest disease
* significant visual or auditory impairment
* parents with limited literacy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of Children with diplegic CP age range 2 to 4.5
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Parental stress | 1 day - one session
  Parental stress will be measured by the Arabic version of the parent stress index-short form (PSI-SF) . PSI-SF is a self-reported questionnaire with 36 items rated on a 5-point Likert scale (strongly agree or strongly disagree). The score of the measure ranged between 36 and 180, and a lower score indicates a better outcome.

SECONDARY OUTCOMES:
Quality of life of parents | 1 day - one session
  Quality of life (QoL) will be measured by the family impact module (PedsQL) and quality-of-life inventory.
Gross motor impairments | 1 day - one session
  Gross motor impairments will be assessed via gross motor classification system

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Privacy Concerns: IPD can be very detailed and contain sensitive information about participants, such as their medical history, diagnoses, and treatment responses. Sharing this data could potentially identify participants, even if it is de-identified. This can be a major concern, especially for studies involving rare diseases or conditions.
  Data Security: Making IPD publicly available raises risks of data breaches or unauthorized access. Researchers need to be confident they have robust security measures in place to protect sensitive participant information.

REFERENCES:
- [Result] Dubois-Comtois K, St-Onge J, St-Laurent D, Cyr C. Paternal distress and child behavior problems in low-SES families: Quality of father-child interactions as mediators. J Fam Psychol. 2021 Sep;35(6):725-734. doi: 10.1037/fam0000830. Epub 2021 Mar 11. PMID 33705176
- [Result] Villamor E, Tedroff K, Peterson M, Johansson S, Neovius M, Petersson G, Cnattingius S. Association Between Maternal Body Mass Index in Early Pregnancy and Incidence of Cerebral Palsy. JAMA. 2017 Mar 7;317(9):925-936. doi: 10.1001/jama.2017.0945. PMID 28267854